CLINICAL TRIAL: NCT00167947
Title: A Randomized, Open Label Study to Evaluate the Effects of a Regimen With Sirolimus,Low Doses Cyclosporine and Steroids vs a Regimen With Sirolimus and Steroids, After an Induction Period With Basiliximab, Sirolimus,Cyclosporine and Steroids in de Novo Renal Transplant Patients.
Brief Title: Study Evaluating Sirolimus in Kidney Transplant Recipients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0468E-101629
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2008-03-14 (Estimated); Status verified 2008-03

CONDITIONS: Kidney Failure; Graft vs Host Disease
Keywords: Kidney; Transplant
MeSH Terms: conditions — Renal Insufficiency; Graft vs Host Disease | interventions — Cyclosporine; Steroids; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Cyclosporine; Drug: Steroids; Drug: Rapamune (Sirolimus)
- B (Experimental)
  Interventions: Drug: Cyclosporine; Drug: Steroids; Drug: Rapamune (Sirolimus)

INTERVENTIONS:
Drug: Cyclosporine — Arm 1= Rapamune+ low dose Cyclosporine+steroids "Arm 2= 1° day rapamune 15 mg/die + steroids 2°-7° day Rapamune 5mg/die + steroids In both arms, Cylcoporine is stopped "
Drug: Steroids — Arm 1= Rapamune+ low dose Cyclosporine+steroids "Arm 2= 1° day rapamune 15 mg/die + steroids 2°-7° day Rapamune 5mg/die + steroids In both arms, Cylcoporine is stopped "
Drug: Rapamune (Sirolimus) — Arm 1= Rapamune+ low dose Cyclosporine+steroids "Arm 2= 1° day rapamune 15 mg/die + steroids 2°-7° day Rapamune 5mg/die + steroids In both arms, Cylcoporine is stopped "

SUMMARY:
Renal function at 12 months assessed by calculated creatinine clearance.

ELIGIBILITY:
Inclusion Criteria:

* Age is older than 18 years.
* End-stage renal disease, with subjects scheduled for kidney transplant.
* Women of childbearing potential must not be pregnant and agree to medically acceptable method of contraception throughout the treatment period and for 3 months following discontinuation of assigned treatment.

Other inclusion applies.

Exclusion Criteria:

* Evidence of active systemic or localized major infection.
* Use of any investigational drug or treatment up to 4 weeks prior to study entry.
* Known hypersensitivity to SRL or its derivatives, macrolide antibiotics, corticosteroids, basiliximab.
* Multiple organ transplants (i.e., prior or concurrent transplantation of any organs other than renal transplant).
* Immunosuppression therapies other than those allowed in the protocol.
* Treatment with voriconazole, terfenadine, cisapride, astemizole, pimozide, or ketoconazole (all known to interact with SRL) that is not discontinued prior to study entry.

Other exclusion applies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2005-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and efficacy of an immunosuppressive regimen using synergic action of SRL and CsA, but which will limit (ab initio), the nephrotic effect of such combination. To compare Rapamune/low dose Cyclosporine vs. Rapamune/Steroids. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Italy, decresg@wyeth.com
Locations (13):
- Italy (13):
  - Rome, Lazio
  - Palermo, Sicily
  - Bari
  - Bologna
  - Cagliari
  - Florence
  - L’Aquila
  - Milan
  - Pisa
  - Sassari
  - Siena
  - Udine
  - Varese